CLINICAL TRIAL: NCT01638208
Title: Spectrum of Gastrointestinal Microbiota in Patients With IBS-D Before and After Treatment With VSL#3.
Brief Title: Changes in Gastrointestinal Microbiota Using VSL#3 in Patients With IBS-D
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Pratap Nitesh, Consultant Gastroenterologist, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIG-VSL#3-IBS-NP
Record Dates: First submitted 2012-07-06; First posted 2012-07-11 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VSL#3 (Experimental): Patients with IBS-D as per ROME III
  Interventions: Drug: VSL#3
- Healthy Controls (No Intervention): Healthy controls

INTERVENTIONS:
Drug: VSL#3 — Dosage Form: Capsules (Details as given below); Dose and duration of treatment: 1 capsule b.i.d for 8 weeks; Each capsule contains 112.5 Billion CFU of the following 8 strains of bacteria, 4 lactobacilli strains (L. acidophilus, L. plantarum, L. paracasei, L. delbrueckii subsp bulgaricus), 3 bifidobacteria strains (B. breve, B. infantis, B. longum) and 1 strain of S. thermophilus).
  Other Names: probiotic
  Arms: VSL#3

SUMMARY:
Aim

To compare changes in gut microbiota of IBS patients and healthy controls using next generation sequencing method like Illumina sequencing based on 16S rDNA profiling.

The major objectives of the study are:

To characterize type of bacterial species and compare diversity of the host's gut microbiota in 20 Irritable bowel syndrome (IBS) patients with 16 healthy controls (HCs) using high through put culture-independent method like Illumina sequencing.

To study modulation of gut microbiota profile after treatment with probiotics (VSL #3) for 8 weeks.

To study the improvement of symptoms after modulation of gut microbiota with probiotics (VSL #3) for more than 8 weeks.

DETAILED DESCRIPTION:
Introduction

The role of the commensal flora in many disease states, including irritable bowel syndrome, inflammatory bowel disease, and even obesity, is now accepted and will undoubtedly lead to new therapeutic strategies. The recently NIH-initiated Human Microbiome Project will allow better understanding of the role of this complex intestinal community in human health and disease. On the clinical side, we are exploring the more common pathogenic bacterial strains in Irritable bowel syndrome patients and use of probiotics in this functional gastrointestinal disease. We are taking support from Genotypic institute, Bangalore for Illumina sequencing facility.

Asian Institute of Gastroenterology, the parent institution, is a 200 bed tertiary care referral hospital providing services to patients with GI diseases, with a daily attendance of 400 out-patients and 200 in-patients. The long term goals of the investigators, involving basic researchers and clinicians, include development of technological resources and applications of biotechnology for use in clinical trials to improve survival rates of patients with GI diseases. The major volume of the outpatient cases comprise of patients with irritable bowel syndrome. Altered GI microbiota may contribute to IBS symptoms and studying dysbiosis in gut microbiota is an important to develop therapy for IBS.

ELIGIBILITY:
Inclusion Criteria:

* Patients satisfying Rome III Criteria

Exclusion Criteria:

* Antimicrobial medication during last 2 months
* Probiotics medication during last 2 months
* Pregnant or lactating patients
* Previous major or complicated abdominal surgery
* Positive test for HIV, HBV or HCV

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-08; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of symptoms after modulation of gut microbiota with probiotic, VSL#3 | 8 wks
  To study modulation of gut microbiota profile after treatment with probiotics (VSL #3) for 8 weeks.

SECONDARY OUTCOMES:
Comparison of GI microbiota before and after treatment | 8 wks
  To characterize type of bacterial species and compare diversity of the host's gut microbiota in 20 Irritable bowel syndrome (IBS) patients with 16 healthy controls (HCs) using high through put culture-independent method like Illumina sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nitesh Pratap, DM, Principal Investigator — Asian Institute of Gastroenterology; Dr. Nageshwar Reddy, DM, Study Director — Asian Institute of Gastroenterology
Locations (1):
- Asian Institute of Gstroenterology, Hyderabad, Andhra Pradesh, India